CLINICAL TRIAL: NCT05187689
Title: Tushirikiane4MH: Mental Health Literacy and Mental Health Promotion With Urban Refugee Youth in Kampala, Uganda
Brief Title: Mental Health Literacy and Mental Health Promotion With Urban Refugee Youth in Kampala, Uganda
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Toronto (Other)
Collaborators: Young African Refugees for Integral Development (Unknown)
Responsible Party: Principal Investigator, Carmen Logie, MSW, PhD, Associate Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 40965
Record Dates: First submitted 2021-12-23; First posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: Mental Health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The two intervention arms will be compared to the control arm of the study using a pre- and post-intervention survey. There will also be a follow-up survey 8 weeks after the study is complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual reality and mental health literacy intervention (Experimental): This arm will participate in an interactive virtual reality experience to learn and practice mental health literacy and psychological first aid skills, supplemented by mhealth SMS with informational bidirectional messages.
  Interventions: Behavioral: VR + MHL intervention
- Group Problem Management+ and VR/mental health literacy (Experimental): This arm will participate in an interactive virtual reality experience to learn and practice mental health literacy and psychological first aid skills, supplemented by mhealth SMS with informational bidirectional messages. This arm will also participate in an 5-week Group Problem Management Plus intervention, a group based problem solving intervention.
  Interventions: Behavioral: Group PM+
- Control (No Intervention): This is a waitlist control. After Arms 1 and 2 are complete, the waitlist will receive the Group Problem Management Plus 5 week intervention on its own.

INTERVENTIONS:
Behavioral: VR + MHL intervention — The intervention will include: 1) a Virtual Reality (VR) interactive and immersive 30-minute session viewed using a low cost VR headset; and 2) an 8-week program of weekly WelTel SMS check-ins managed by Peer Navigators (PNs), weekly WelTel SMS blasts informed by Psychological First Aid (PFA) with mental health literacy (MHL) messages developed with PN, and weekly WelTel web-based secure platform social group discussions on MHL, stress coping, and stigma moderated by PN alongside a trained Coordinator. Weekly MHL WelTel platform moderated discussion foci will address MHL, stigma and stress coping strategies, including self-compassion and other strategies that emerge from the urban refugee youth interviews and focus groups, through diverse methods, including: 'scenarios' mimicking real life situations; a 'question box'; sharing photos demonstrating stress coping strategies; memes; songs; and ways participants interrupted stigma in their daily lives.
  Arms: Virtual reality and mental health literacy intervention
Behavioral: Group PM+ — Participants will attend small groups (5-6 participants with a PN and a coordinator supporting) outdoors with physically distancing, for Group PM+ sessions following the adapted WHO Group-PM+ manual (adaptations made in Phase 1 explain above) 5 weekly 3-hour sessions delivered by PN who will co-facilitate sessions with the Coordinator. Each session has a mechanism of action:
  1. Managing stress: mechanism of action-identify goals, learn deep breathing and techniques for stress management
  2. Managing problems: mechanism of action-identify 1 solvable practical problem, brainstorm possible solutions together
  3. Get going, keep doing: mechanism of action-learn about depression and inactivity, identify and plan small enjoyable activities
  4. Strengthen social support: mechanism of action-discuss a range of social support resources, make plan to increase social support
  5. Staying well: mechanism of action- this session reviews all of the mechanisms of action in the prior 4 sessions
  Arms: Group Problem Management+ and VR/mental health literacy

SUMMARY:
From our previous studies, we know that urban refugee youth commonly report depressive symptoms. The primary aim of this study is to compare the effectiveness of youth-tailored interventions to improve mental health literacy and reduce mental health stigma among urban refugee youth in Kampala, Uganda. There will be two intervention arms and one control arm. The first intervention arm will involve a VR experience that focuses on mental health literacy and coping strategies, as well as SMS check-ins from peer navigators (PN) trained in psychological first aid. The second intervention arm will involve an adapted version of the WHO's Group Problem Management Plus. The primary outcomes are to a) increase mental health literacy (knowledge and understanding of mental health generally and of specific disorders; b) increase attitudes towards mental health help-seeking, c) reduce depression, d) increase adaptive coping strategies; e) reduce mental health stigma, f) improve mental wellbeing, and g) increase level of functioning. Participants will complete a pre- and post-intervention survey as well as a follow-up survey.

ELIGIBILITY:
Inclusion Criteria:

1. living in one of the 5 informal settlements in Kampala we already work with (Nsambya, Katwe, Rubaga, Kabalagala, Kansanga);
2. self identify as a woman or man (transgender inclusive);
3. identify as a refugee/displaced person/having refugee parents;
4. aged 16-25;
5. own a mobile phone;
6. speak Swahili, Luganda, Kirundi, Kinyarwanda, French or English and can provide informed consent.

Exclusion Criteria:

-

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 330 (Estimated)
Dates: Start 2022-01-31 (Estimated); Primary Completion 2022-05-27 (Estimated); Study Completion 2022-05-27 (Estimated)

PRIMARY OUTCOMES:
Mental health literacy | change from baseline at 16 weeks
  Measured using a modified depression literacy scale validated in Low- and Middle- Income Countries (LMICs)
Attitudes towards mental health help seeking | change from baseline at 16 weeks
  Measured using the Inventory of Attitudes towards Seeking Mental Health Services
Depression | change from baseline at 16 weeks
  Measured using the PHQ-9
Adaptive coping strategies | change from baseline at 16 weeks
  Measured by the Kidcope and Self-Compassion Scale for Youth
Mental Health Stigma | change from baseline at 16 weeks
  Measured using the Brief Version of the Internalized Stigma of Mental Illness (ISMI) Scale
Mental wellbeing | change from baseline at 16 weeks
  Measured using the WHO-Five Wellbeing Scale
Level of functioning | change from baseline at 16 weeks
  Measured usingWHO Disability Assessment Schedule

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Logie, PhD, Principal Investigator — University of Toronto

IPD SHARING:
Plan to Share IPD: Yes
The final deidentified data set will be available to users who enter a data-sharing agreement with us. Users will need to (1) secure ethics approval from both their institution and the University of Toronto research ethics board; (2) commit to use the data solely for research purposes, and not to identify any individual participant; (3) commit to securing the data using the appropriate computer technology such as encryption; and (4) commit to destroying or returning the data after analyses are complete.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will become available 12 months after study completion.
Access Criteria: The final deidentified data set will be available to users who enter a data-sharing agreement with us. Users will need to (1) secure ethics approval from both their institution and the University of Toronto research ethics board; (2) commit to use the data solely for research purposes, and not to identify any individual participant; (3) commit to securing the data using the appropriate computer technology such as encryption; and (4) commit to destroying or returning the data after analyses are complete.

REFERENCES:
- [Derived] Logie CH, Okumu M, Kortenaar JL, Gittings L, Khan N, Hakiza R, Kibuuka Musoke D, Nakitende A, Katisi B, Kyambadde P, Khan T, Lester R, Mbuagbaw L. Mobile Health-Supported Virtual Reality and Group Problem Management Plus: Protocol for a Cluster Randomized Trial Among Urban Refugee and Displaced Youth in Kampala, Uganda (Tushirikiane4MH, Supporting Each Other for Mental Health). JMIR Res Protoc. 2022 Dec 8;11(12):e42342. doi: 10.2196/42342. PMID 36480274